CLINICAL TRIAL: NCT01862198
Title: Pilot Study on the Usefulness of Endoscopic Ultrasound-guided Biliary Drainage With a Newly Designed Hybrid Metallic Stent
Brief Title: The Usefulness of Endoscopic Ultrasound-guided Biliary Drainage With a Newly Designed Hybrid Metallic Stent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Tea Jun Song, Assistant professor, Inje University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2012-1819-0002
Record Dates: First submitted 2013-05-19; First posted 2013-05-24 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Bile Duct Obstruction; Disorder of Bile Duct Stent; Neoplasms
MeSH Terms: conditions — Cholestasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hybrid metallic stent (Experimental): Patients group who were inserted a hybrid metallic stent
  Interventions: Device: EUS-guided biliary drainage with a hybrid metallic stent

INTERVENTIONS:
Device: EUS-guided biliary drainage with a hybrid metallic stent — EUS-guided biliary drainage with a newly designed hybrid metallic stent

SUMMARY:
The purpose of this study is to investigate the feasibility and safety of endoscopic ultrasound-guided biliary drainage with a newly designed hybrid metallic stent.

DETAILED DESCRIPTION:
Endoscopic ultrasound-guided biliary drainage with a fully covered metallic stent was a safe and effective method in patients with malignant biliary obstructions and had a comparatively long patency duration. Nevertheless, the significant rate of distal stent migration cannot be ignored, suggesting the need for a newly designed metallic stent for endoscopic ultrasound-guided biliary drainage.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* The presence of an unresectable malignant biliary obstruction
* Failed conventional ERCP stenting

Exclusion Criteria:

* Age < 20 years
* An inability to sedate the patient due to advanced heart or pulmonary diseases
* A lack of informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The stent patency rate | Up to 48 weeks

SECONDARY OUTCOMES:
Patients' survival rate | Up to 48 weeks
Complication rate related to the hybrid stents | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Soo Lee, MD, PhD, Study Chair — Department of Internal Medicine, University of Ulsan College of Medicine, Asan Medical Center, Seoul , South Korea
Locations (2):
- South Korea (2):
  - Inje University Ilsan Paik Hospital, Koyang
  - Asan Medical Center, Seoul